CLINICAL TRIAL: NCT00828191
Title: Efficacy and Tolerability of Subcutaneous Progesterone (IBSA) Versus Vaginal Progesterone for Luteal Phase Support in Patients Undergoing In Vitro Fertilization (IVF)
Brief Title: Subcutaneous Progesterone Versus Vaginal Progesterone Tablets for Luteal Phase Support in In Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07USA/Prg05
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2012-12-26 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: In Vitro Fertilization
Keywords: Luteal support in IVF
MeSH Terms: interventions — Progesterone

ARMS (2):
- Progesterone SC (Experimental)
  Interventions: Drug: Progesterone
- Progesterone Tablets (Active Comparator)
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — 25 mg, once a day, SC
  Arms: Progesterone SC
Drug: Progesterone — 100 mg, twice a day, vaginally
  Arms: Progesterone Tablets

SUMMARY:
Prospective, open, randomized, parallel, multicenter, two-arm trial to evaluate the efficacy and tolerability of a new progesterone formulation to be used for luteal support in IVF (Progesterone-IBSA) administered subcutaneously at a daily dose of 25 mg versus Progesterone tablets administered intravaginally at 100 mg twice daily for a total dose of 200 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent;
* BMI < 30 kg/m2;
* Age 18 - 42 (upon starting COH);
* <3 prior ART cycles (IVF, ICSI and related procedures);
* Baseline (day 2-3 of cycling) FSH <15 IU/L and E2 <80 pg/mL;
* Normal uterine cavity as per recent hysterosalpingogram, sonohysterogram or hysteroscopic exam (i.e. no polyps or protruding submucosal fibroids);
* Patients must have at least three retrieved oocytes.

Exclusion Criteria:

* Intramural uterine fibroids that distort the uterine cavity or polyps >1 cm;
* Stage III or IV endometriosis (no endometriomas);
* Hydrosalpinges;
* History of past poor response to COH resulting in canceling ART;
* Use of thawed/donated oocytes;
* Use of thawed/donated embryos;
* Gestational carrier;
* Patients affected by pathologies associated with any contraindication of being pregnant;
* Hypersensitivity to study medication;
* Uncontrolled adrenal or thyroid dysfunction;
* History of conditions (i.e. toxic shock syndrome) that would contraindicate use of a vaginal progesterone product;
* History of arterial disease;
* Patients with hepatic impairment (liver function tests > 2x upper limits of normal);
* Patients with dermatologic disease;
* Patients with renal impairment (estimated creatinine clearance <60 mL/min/1.73 m2);
* Neoplasias (current) or history of neoplasia that may be responsive to progesterone;
* High grade cervical dysplasia;
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages, wherein pregnancy developed to a minimum of a gestational sac on TVUS;
* Participation in a concurrent clinical trial or in another trial within the past 2 months;
* Use of concomitant medications that might interfere with the study evaluation;
* Pre-implantation genetic diagnosis/screening

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Reproductive Partners Medical Group, Inc., Redondo Beach, California
  - Fertility Physicians of Northern California, San Jose, California
  - Stanford University Medical Center, Stanford, California
  - Fertility and Surgical Associates of California, Thousand Oaks, California
  - Center for Reproductive Medicine, Orlando, Florida
  - Idaho Center for Reproductive Medicine, Boise, Idaho
  - Center for Assisted Reproduction, Bedford, Texas
  - Seattle Reproductive Medicine, Seattle, Washington

REFERENCES:
- [Derived] Griesinger G, Trevisan S, Cometti B. Endometrial thickness on the day of embryo transfer is a poor predictor of IVF treatment outcome. Hum Reprod Open. 2018 Jan 29;2018(1):hox031. doi: 10.1093/hropen/hox031. eCollection 2018. PMID 30895243
- [Derived] Baker VL, Jones CA, Doody K, Foulk R, Yee B, Adamson GD, Cometti B, DeVane G, Hubert G, Trevisan S, Hoehler F, Jones C, Soules M. A randomized, controlled trial comparing the efficacy and safety of aqueous subcutaneous progesterone with vaginal progesterone for luteal phase support of in vitro fertilization. Hum Reprod. 2014 Oct 10;29(10):2212-20. doi: 10.1093/humrep/deu194. Epub 2014 Aug 6. PMID 25100106

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone SC: Progesterone SC given at a daily dose of 25 mg.
- Progesterone Tablets: Progesterone vaginal tables 100 mg given twice à day.
Period: Overall Study
Arm/Group | Progesterone SC | Progesterone Tablets
Started | 400 (Randomized patients) | 400 (Randomized patients)
Completed | 392 (Patients with at least one embryo transferred.) | 390 (Patients with at least one embryo transferred.)
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone SC | Progesterone Tablets | Total
Number analyzed (Participants) | 400 | 400 | 800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 400 | 400 | 800
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (4.4) | 34.3 (4.5) | 34.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400 | 400 | 800
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 400 | 400 | 800

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Time Frame: 10 weeks after treatment start
Population: All randomized patients were included in the analysis
Measure: Number; unit: percentage of randomized patients
Arm/Group | Progesterone SC | Progesterone Tablets
Number analyzed (Participants) | 400 | 400
percentage of randomized patients | 40.8 | 43.3
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Tablets; The non -inferiority hypothesis to be tested for the primary endpoint was that the ongoing pregnancy rate (oPR) in the test group (Pe)was lower than the oPR in the control group (Pc)against the alternative one that the oPR in the test group was equal to or higher than the oPR in the control group. H0 : Pc>= Pe + d(-10%) H1 : Pc< Pe + d(-10%); Test type: Non-Inferiority or Equivalence — The null hypothesis (H0) was tested against the alternative by calculating a two-sided 95% confidence interval for the difference in ongoing pregnancy rates. If the lower bound of the 95% confidence interval was greater than the non-inferiority limit (-10.0%), the null hypothesis was rejected and the test group considered not inferior to the control treatment; p = 0.52, Fisher Exact; Difference in pregnancy rates = -2.5, 95% CI 2-sided [-9.4 to 4.4]

2. Secondary Outcome: Implantation Rate
Description: Implantation rate was defined as the number of gestational sacs divided by the number of embryos transferred (%). This value was calculated for all the patients who had at least one embryo transferred.
Time Frame: 4-5 weeks after treatment start
Population: Patient who had at least one embryo transferred.
Measure: Mean (Standard Deviation); unit: percentage of embryos transferred
Arm/Group | Progesterone SC | Progesterone Tablets
Number analyzed (Participants) | 392 | 390
percentage of embryos transferred | 33.2 (42.0) | 35.1 (40.9)
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Tablets; Test type: Superiority or Other; p = 0.54, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.6 to 4.0], Standard Error of Mean 1.48

3. Secondary Outcome: Delivery Rate
Time Frame: nearly 9 months after treatment start
Population: All randomized patients
Measure: Number; unit: percentage of randomized patients
Arm/Group | Progesterone SC | Progesterone Tablets
Number analyzed (Participants) | 400 | 400
percentage of randomized patients | 40.5 | 42.5
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Tablets; Test type: Superiority or Other; p = 0.62, Fisher Exact; Risk Difference (RD) = -2.0, 95% CI 2-sided [-8.8 to 4.8]

ADVERSE EVENTS:
Description: None of the patients reported SAE considered as related to study drugs.
Arm/Group | Progesterone SC | Progesterone Tablets
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/400
Other Adverse Events (participants affected / at risk) | 156/400 | 161/400
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone SC (N=400) | Progesterone Tablets (N=400)
Injection site bruising (General disorders) | 37 (38) | 0 (0)
Injection site discomfort (General disorders) | 57 (68) | 0 (0)
Vaginal discharge (General disorders) | 0 (0) | 50 (50) — AE associated with vaginal administration
Abdominal discomfort (Gastrointestinal disorders) | 21 (25) | 28 (35)
Constipation (Gastrointestinal disorders) | 12 (13) | 23 (23)
Headache (Nervous system disorders) | 28 (31) | 36 (37)
Breast pain/tenderness (Reproductive system and breast disorders) | 17 (17) | 42 (44)
vaginal hemorrage (Reproductive system and breast disorders) | 28 (30) | 30 (34)

LIMITATIONS AND CAVEATS:
No limitations of the trial reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No